CLINICAL TRIAL: NCT02962297
Title: VENS is a Multicenter, Randomized, Double-masked, Placebo Parallel Controlled Trial to Evaluate the Efficacy and Safety of Treatment With Vitamin E Softgel in Non Diabetic Adults With NASH Compared to Treatment With Placebo in China
Brief Title: Vitamin E Versus Placebo for the Treatment of Non Diabetic Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Medicine Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry); The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VENS
Record Dates: First submitted 2016-10-27; First posted 2016-11-11 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2020-11

CONDITIONS: NASH (Non-Alcoholic Steatohepatitis)
Keywords: Vitamin E, Non Diabetic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- treatment group (Experimental): Vitamin E softgel,100mg,Tid,orally, 96 weeks. All participants receive standardized recommendations for life-style modification (Diet modification, weight loss, exercise).
  Interventions: Drug: Vitamin E softgel
- placebo group (Placebo Comparator): A similar appearing placebo softgel , Vitamin E -Placebo, Tid, orally, 96 weeks, All participants receive standardized recommendations for life-style modification (Diet modification, weight loss, exercise).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin E softgel — All participants receive standardized recommendations for life-style modification (Diet modification, weight loss, exercise).
  Arms: treatment group
Drug: Placebo — All participants receive standardized recommendations for life-style modification (Diet modification, weight loss, exercise).
  Height and weight, waist-to-hip ratio Review of diet and exercise
  Arms: placebo group

SUMMARY:
VENS is a multicenter, randomized, double-masked, placebo parallel controlled trial to evaluate the efficacy and safety of treatment with vitamin E softgel in non diabetic adults with NASH compared to treatment with placebo in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 -75, no limitation for ethnic and gender
2. Body Mass Index(BMI) < 35 kg/m2
3. Patients with nonalcoholic steatohepatitis (NASH) based on liver biopsy obtained within 6 months before randomization. The histological evidence of NASH was defined as Non - alcoholic fatty liver disease activity score（NAS）≥ 4 (according to Nonalcoholic Steatohepatitis Clinical Research Network, NASH CRN) with a minimum 1 score for steatosis, lobular inflammation, and hepatocyte ballooning respectively.
4. Fibrosis stage 0-3 according to nonalcoholic steatohepatitis clinical research network（NASH CRN).
5. Without history of significant alcohol consumption for a period of more than 3 months within 5 years (<10 g/day for female and < 20 g/day for male).
6. The lab test results should meet the requirements:

   ① Alanine aminotransferase （ALT） < 5 times of normal upper limit

   ② Creatinine (Cr)< normal upper limit

   ③ Albumin （ALB）> 3.5g/L

   ④ International normalized ratio（INR）= 0.8-1.3

   ⑤ Fasting plasma glucose(FPG) < 126mg/dL（7mmol/L） and/or 2h postprandial plasma glucose (PPG) < 200mg/dL（11.1mmol/L）and/ or HbA1C < 6.5 %
7. If a participant with hypertension, he/she was required a stable antihypertensive drug(s) to keep blood pressure stable.(blood pressure < 140/90 mmHg) 3 months prior to randomization.
8. If a participant using a statin or fibrate, he/she was required on a stable dose to keep lipid stable (triglyceride(TG) < 1.7 mmol/L, total cholesterol (TC) < 5.72 mmol/L, LDL-c < 3.64 mmol/L) 3 months prior to randomization.
9. Women of childbearing potential: negative pregnancy test during screening or at randomization or willingness to use an effective form of birth control during the trial(at least include one barrier contraceptive method) and not breast feeding
10. Men must agree to use an effective form of birth control during the trial(at least include one barrier contraceptive method)
11. All participants are needed to sign the informed consent form.

Exclusion Criteria:

1. Evidence of other form of acute or chronic liver disease. (Virus hepatitis, Hereditary hemochromatosis, Hepatolenticular degeneration, Alcoholic liver disease, Drug-induced hepatopathy).
2. History of diabetic mellitus or use of antidiabetic drugs.
3. Known heart failure of New York Heart Association class 2, 3, or 4.
4. Wear of cardiac pacemaker.
5. Hypothyroidism (TSH > 2 times of upper normal limit).
6. History of disease affecting drug absorption, distribution, metabolism (inflammatory bowel disease, gastrointestinal surgery, chronic pancreatitis, gluten allergy, vagotomy).
7. Use of anti-NASH drugs within 3 months before randomization (metformin, thiazolidinediones, dipeptidyl peptidase-4 (DPP-4) inhibitor, glucagon-like peptide-1(GLP-1), sodium glucose contransporter2(SGLT2), S-adenosylmethionine -e(SAM-e), polyene phosphatidyl choline, glycyrrhizin, bicyclol, reduced glutathione, betaine, fish oil, silymarin,oberbic acid/ursodeoxycholic acid (OCA/UDCA), phosphodiesterase (PDE)-inhibitor, gemfibrozil, vitamin E, long term antibiotic (>1 week).
8. Positivity of antibody to Human Immunodeficiency Virus.
9. Inability to safely obtain liver biopsy.
10. Known intolerance to vitamin E
11. Inability to fill out diary card, to manage diet and exercise, poor compliance.
12. Dependence or abuse of alcohol and/or drugs.
13. Any other condition which in the opinion of investigator would impede compliance or hinder completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Improvement in hepatic histology | after 96 weeks of treatment
  Improvement in hepatic histology after 96 weeks of treatment as determined by liver biopsies compared to baseline. (Independent pathological evaluation committee was charged with interpreting of the histological characteristic and that allows for assessment of changes with therapy). The definition of histologic improvement requires all three of the following criteria: ① either improvement in NAS by at least 2 points or post-treatment NAS of 3 points or less, ② at least 1 point improvement in the score for ballooning or lobular inflammation③ no worsening of fibrosis stages.

CONTACTS AND LOCATIONS:
Overall Officials: Junping Shi, Phd, Principal Investigator — The Affiliated Hospital of Hangzhou Normal University
Locations (15):
- China (15):
  - Beijing Ditan Hospital Capital Medical University, Beijin, Beijing Municipality
  - 302 Military Hospital of China, Beijing
  - Beijing YouAn Hospital Capital Medical Univercity, Beijing
  - West China Hospital, Sichuan university, Chengdu
  - The first Affiliated Hospital, Sun Yat-sen University, Guangdong
  - Guangdong Provincial Chinese Medicine Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Southwest Medical University Affiliated, Luzhou
  - The Second Hospital of Nanjing, Nanjing
  - The First Hospital of China Medical University, Shenyang
  - The second people's Hospital of Tianjin, Tianjin
  - The First Affiliated Hospital of Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhu
  - General Hospital Ningxia Medical, Yinchuan

REFERENCES:
- [Derived] Song Y, Ni W, Zheng M, Sheng H, Wang J, Xie S, Yang Y, Chi X, Chen J, He F, Fan X, Mi Y, Zhang J, Wang B, Bai L, Xie W, Zhong B, Yeo YH, Rui F, Zang S, Li J, Shi J; Chinese NAFLD Clinical Research Network (CNAFLD CRN). Vitamin E (300 mg) in the treatment of MASH: A multi-center, randomized, double-blind, placebo-controlled study. Cell Rep Med. 2025 Feb 18;6(2):101939. doi: 10.1016/j.xcrm.2025.101939. PMID 39970876
- [Derived] Zang S, Chen J, Song Y, Bai L, Chen J, Chi X, He F, Sheng H, Wang J, Xie S, Xie W, Yang Y, Zhang J, Zheng M, Zou Z, Wang B, Shi J; Chinese NAFLD Clinical Research Network (CNAFLD CRN). Haptoglobin Genotype and Vitamin E Versus Placebo for the Treatment of Nondiabetic Patients with Nonalcoholic Steatohepatitis in China: A Multicenter, Randomized, Placebo-Controlled Trial Design. Adv Ther. 2018 Feb;35(2):218-231. doi: 10.1007/s12325-018-0670-8. Epub 2018 Feb 6. PMID 29411270